CLINICAL TRIAL: NCT00812721
Title: Tears Substitutions and Their Effects on Higher Order Aberrometery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Gina Rogers (Other)
Responsible Party: Sponsor-Investigator, Gina Rogers, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Iowa RR 01
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye Syndrome
Keywords: higher order aberrations; tear blur
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Placebo Comparator): Preservative Free Saline
  Interventions: Other: Preservative Free Saline
- 2 (Active Comparator): Optive (TM)
  Interventions: Other: Optive
- 3 (Active Comparator): Refresh Moderate/Severe (TM)
  Interventions: Other: Refresh Moderate/Severe
- 4 (Active Comparator): Systane (TM)
  Interventions: Other: Systane
- 5 (Active Comparator): Systane Ultra (TM)
  Interventions: Other: Systane Ultra

INTERVENTIONS:
Other: Preservative Free Saline — One drop will be instilled into each eye once
  Arms: 1
Other: Optive — One drop will be instilled into each eye once
  Arms: 2
Other: Refresh Moderate/Severe — One drop will be instilled into each eye once
  Arms: 3
Other: Systane — One drop will be instilled into each eye once
  Arms: 4
Other: Systane Ultra — One drop will be instilled into each eye once
  Arms: 5

SUMMARY:
Hypothesis is that tear substitutions cause blur after they are instilled. The investigators will use aberrometry as a measurement over time after a tear formulation is used and try to determine if there are any measurable change in higher order aberrations between different tear formulations and how long it takes to return to pre-instillation measurements thus providing information on duration of the tear drop. 4 commercially available "dry eye" artificial tears formulations will be used and preservative saline will act as a control. The study will be conducted on subjects that do not have clinical evidence of dry eye syndrome to focus the data on the blur effects of the tear substitutions.

DETAILED DESCRIPTION:
Once consent is obtained the subject will choose from available time slots. Each subject will come to the UIHC Department of Ophthalmology at designated times for approximately one hour on five different days, for a total time commitment of approximately 5 hours. Each subject will receive the same 4 artificial tear substitutes and saline, one different drop each day. One of the four tear substitutes (brands: Systane, Systane Ultra, Optive, and Refresh) will be tested on each of the days. One drop will be used each day and the protocol of each day will be the same, the only factor changing from day to day is the drop that is being evaluated. On each study day, the subject will have a pre-instillation measurement of their higher order aberrometry of each eye. One drop of the designated drop will be placed into each of the eyes. Subsequent aberrometry measurements of each eye will be taken at immediately post-instillation, 5 minutes, 30 minutes and 60 minutes post instillation. The same protocol will be followed with a saline drop and thus each patient will act as a control.

There is no long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that do not have any complaints of dry eye and confirmed by ocular surface disease index questionnaire.
* Visually correctable to 20/20 in each eye.
* Non contact lens wearer.
* No history of systemic disease associated with dry eye syndromes.
* No current use of ocular medications.
* Adult volunteers who agree to HIPAA standards and sign informed consent.

Exclusion Criteria

* Patients that have dry eye symptoms or slitlamp findings consistent with dry eye.
* Have a systemic condition that is associated with dry eye syndromes.
* Take systemic medications that have dry as a side effect
* Currently use artificial tears.
* Currently are using ocular medications.
* Currently wear contact lenses.
* Enrollment of the investigator's office staff, relatives, or members of their respective households.
* Enrollment of more than one member of the same household.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of a subject's higher order aberrations over time is the primary outcome measure | pre drop instillation, 1, 5, 15, 30, and 60 minutes post instillation

CONTACTS AND LOCATIONS:
Overall Officials: Gina M Rogers, MD, Principal Investigator — University of Iowa Department of Ophthalmology and Visual Sciences; Christine Sindt, OD, Study Director — niversity of Iowa Department of Ophthalmology and Visual Sciences
Locations (1):
- University of Iowa Department of Ophthalmology and Visual Sciences, Iowa City, Iowa, United States